CLINICAL TRIAL: NCT02961023
Title: The Effect of Adding Exercise Training to Optimal Therapy in Pulmonary Arterial Hypertension
Brief Title: The Effect of Adding Exercise Training to Optimal Therapy in PAH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Health Service, United Kingdom (Other Government)
Responsible Party: Principal Investigator, Martin Johnson, Dr Martin K Johnson, National Health Service, United Kingdom
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15/CARD/21, REC 15-WS-197
Record Dates: First submitted 2016-11-08; First posted 2016-11-10 (Estimated); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — Exercise Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Training (Active Comparator): 15 patients are randomised to receive 15 weeks exercise therapy as per study protocol at point of study entry.
  Interventions: Other: Exercise therapy
- Control (Other): 15 patients are randomised to receive 15 weeks of standard care, acting as a control arm, followed by 15 weeks of exercise therapy.
  Interventions: Other: Exercise therapy

INTERVENTIONS:
Other: Exercise therapy — 3-week residential phase and 12-week outpatient phase.
  Residential phase
  * Exercise will be supervised by a physiotherapist and prescribed based on cardiopulmonary exercise testing.
  * A monitored daily program of exercise involving bicycle ergometry, walking, breathing exercises, dumbbell exercises 5 days per week.
  * 1.5 to 2 hours of exercise will be performed daily, with rest intervals.
  * At weekends, lower intensity, unsupervised exercise mirroring the outpatient phase
  * Ongoing exercise prescription will be based on tolerability, progress and HR
  Outpatient phase
  * A training manual will be compiled based on the subjects exercise performance during the residential program and tailored specifically to their needs
  * Participants will be provided with a cycle ergometer, weights and a HR monitor
  * Weekly telephone contact will be made by the study doctor or physiotherapist, with adjustments made to training prescription as necessary

SUMMARY:
Exercise capacity (EC) is limited in pulmonary arterial hypertension (PAH) by impaired right ventricular (RV) function and inability to increase stroke volume (SV). Disease targeted therapy, increases EC by improving SV. Additional factors may contribute to exercise limitation:

* Peripheral and respiratory muscle dysfunction
* Autonomic dysfunction
* An altered profile of inflammation
* Mitochondrial dysfunction.

The enhancement of EC achieved pharmacologically may therefore be limited. Exercise training in PAH improves EC and quality of life (QOL). The changes in physiology responsible for this improvement are not clear. Patients with PAH stable on optimal oral therapy, but not meeting treatment goals, will be enrolled in a 30-week randomised exercise training program.

One arm will undertake training for 15 weeks (3 weeks residential, 12 outpatient), the other will receive standard care for 15 weeks then 15 weeks training.

Aims:

1. Demonstrate that exercise training can enhance EC and QOL when added to optimal drug therapy a UK PAH population.
2. Explore mechanisms of exercise limitation and factors that improve with training, assessing:

   * Cardiac function
   * Skeletal muscle function
   * Autonomic function
   * Respiratory muscle strength
   * Serum and muscle profile of inflammation

Primary outcomes (15 weeks)

1. 6 minute walk distance
2. QOL
3. RV ejection fraction

DETAILED DESCRIPTION:
Pulmonary arterial hypertension (PAH) is characterised by increased pulmonary vascular resistance (PVR) and elevation of pulmonary artery pressure (PAP) at rest, which rises markedly on exercise. Traditionally, exercise limitation had been attributed to impaired right ventricular (RV) function and an inability of the heart to increase stroke volume (SV) in response to exercise. Disease targeted therapy improves SV by reducing PVR and therefore afterload, with combination therapy being superior in this regard. Despite advances in medical therapy, most patients remain symptomatic on treatment. The 2014 UK PAH national audit demonstrates a 65% failure rate of monotherapy at 2 years. This lack of improvement in exercise tolerance suggests additional mechanisms other than poor SV are responsible for exercise limitation. There is consequently a need for new treatment strategies to improve morbidity and mortality in PAH.

Over the past decade, it has been demonstrated that exercise training in PAH can improve exercise capacity and quality of life (QOL). Exercise training has been shown to result in more significant improvements in exercise capacity and QOL than the majority of pharmacological therapies, with reassuring safety and health economics. Currently, exercise therapy is not part of standard care in the UK and many other European countries. There are several unanswered questions that pose a barrier to its widespread implementation; these fall into three main domains:

A. Relationship with drug therapy

The standard of PAH care is moving towards combination therapy. In the previous studies assessing the effect of exercise therapy, over half of patients have been on monotherapy. No study has exclusively assessed the effect of exercise training in addition to optimal PAH therapy.

B. Health care setting

The strongest supporting evidence for exercise training as an effective therapy in PAH originates from a single centre in Germany, where there are long established, dedicated cardiopulmonary rehabilitation hospitals. These facilities do not exist in many other countries including the UK. It is unclear whether these results can be replicated outwith this robust rehabilitation infrastructure. Data from other centres utilising existing, less intensive outpatient rehabilitation programmes show less certain benefits

C. Mechanistic information

Limited data exist to explain the beneficial effects of exercise training in PAH. There are a number of pathophysiological and pathobiological processes in PAH that may impair the exercise response. These factors have not been studied in relation to the effect of exercise training. In order to best prescribe a PAH specific training programme, it is essential that the underlying mechanisms of improved exercise capacity are fully understood; this will dictate the content, duration and intensity of exercise. It is likely that it affects some or all of the factors listed below:

1. Peripheral muscle structural and functional changes

   In idiopathic PAH (IPAH), there is a reduction in peripheral skeletal muscle capillarisation, oxidative enzyme capacity, shift in type I to II fibres, a higher potential for anaerobic capacity compared with aerobic capacity and reduced function and numbers of mitochondria. Importantly, these changes correlate with exercise capacity and are independent of the severity of pulmonary haemodynamics, suggesting a mechanism other than the atrophying affect of low cardiac output.
2. Autonomic dysfunction

   A higher resting heart rate (HR), reduced heart rate recovery (HRR), reduced HR variability (HRV) and evidence of altered baroreceptor sensitivity (BRS) support autonomic dysfunction in PAH. These findings are independent of haemodynamic severity but correlate with peak oxygen uptake (VO2)
3. Respiratory muscle strength

   Inspiratory and expiratory muscle strength are reduced in IPAH, independently of haemodynamic severity, leading to a reduced ventilatory capacity. Specific respiratory muscle training has been shown to be an important component in exercise training programmes.
4. Direct myocardial effect

   In animal models, exercise training reduces RV hypertrophy and pulmonary artery remodelling, suggesting a direct effect on the pulmonary vasculature and myocardium. Exercise training in patients with stable PH on treatment improved cardiac index and reduced mPAP. In rats with stable monocrotaline induced PAH, exercise trained rats had increased capillary density in cardiomyocytes and improved exercise endurance compared with sedentary matched controls.
5. Micro-RNAs (miRs)

   Systemic angiogenic defects contribute to skeletal muscle microcirculation rarefaction and exercise intolerance, independently of haemodynamic severity. Reduction in the expression of pro-angiogenic miR-126 in the skeletal muscle of humans with PAH correlates with capillary density and peak VO2 and is significantly reduced compared with healthy controls. In a PAH rat model, miR126 down regulation reduces capillary density and this correlates with exercise capacity. In health, change in expression of miRs such as miR-20a correlate with changes in VO2 following exercise training.
6. Cytokines

Inflammatory cytokines may contribute to proteolysis and damage contractile proteins involved in skeletal muscle function. Cytokines such as interleukin (IL)-6, IL-8, IP-10 and monokine induced interferon-γ (MIG) are elevated in the serum of IPAH patients. In chronic thromboembolic pulmonary hypertension (CTEPH), IP-10 negatively correlates with cardiac index and 6mwd. In left ventricular failure, cytokines such as TNF-alpha reduce with exercise training and correlate with improved exercise capacity.

Currently no PAH specific exercise rehabilitation programme exists in the UK. A survey of patient willingness to participate in a program mirroring the successful protocol used in Germany was conducted at the Scottish National Centre for Pulmonary Hypertension. 224 patients with PAH who matched the inclusion criteria of Grunig et al were contacted. 43% (97/224) responded to the survey, 61.9% (60/97) were interested in all components of the rehabilitation program. A further 11.3% (11/97) were interested in outpatient rehabilitation only. It is highly likely that such a program would be of benefit to the PAH population given the demand for it.

Aims

1. Demonstrate that exercise training can enhance exercise capacity and QOL when undertaken in addition to optimal therapy in PAH in a UK setting.
2. Determine the mechanisms of exercise limitation and the factors that improve with training, assessing:

   i. Cardiac function ii. Peripheral muscle structure and function iii. Autonomic function iv. Respiratory muscle strength v. Inflammatory cytokines and miRNA

Original hypothesis

1. Supervised exercise training in patients with stable PAH improves exercise capacity, quality of life and right ventricular ejection fraction. This change occurs through improved RV function, enhanced skeletal and respiratory muscle strength and function and is associated with improvements in autonomic response.
2. Exercise training affects the control mechanisms for skeletal muscle structure and function. Improvements are due to changes in the inflammatory cytokine profile and in expression of miRs associated with angiogenesis, myogenesis and inflammation.

ELIGIBILITY:
Inclusion criteria:

* World health organisation functional class (WHO-FC) II-III
* Stable on optimal disease targeted therapy for ≥ 3 months
* 18 years of age or older

Exclusion criteria

* Unable to provide informed consent
* Significant peripheral vascular disease, neurological or musculoskeletal comorbidity
* Exercise induced syncope, cardiac arrhythmia or chest pain
* Pregnancy
* Specific component exclusions: Cardiac MRI (CMR): Any contraindication to MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-02; Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
6 minute walk distance | 15 weeks
  Change in distance walked in 6 minutes from baseline following 15 weeks of exercise therapy
Quality of life | 15 weeks
  Change in pulmonary hypertension specific (EMPHASIS and CAMPHOR) and generic (SF-36 v2) quality of life scores from baseline to 15 weeks following exercise therapy.
Right Ventricular Ejection Fraction | 15 weeks
  Change in right ventricular ejection fraction from baseline to 15 weeks as measured by cardiac magnetic resonance imaging.

SECONDARY OUTCOMES:
Peak oxygen uptake | 15 weeks
  Peak oxygen uptake as measured by standard incremental cardiopulmonary exercise testing (CPET) at 15 weeks in addition to all other standard CPET variables
Muscle strength and endurance | 15 weeks
  change in quadriceps strength and endurance, and hand grip endurance and strength from baseline to 15 weeks, as measured by a myometer
Transfer factor for lung carbon monoxide | 3 weeks
  Transfer factor for lung carbon monoxide as measured during standard pulmonary function testing. Change from baseline to 3 weeks.
Respiratory muscle strength | 3 weeks
  change maximum inspiratory and maximum expiratory pressure measured following 3 weeks of exercise therapy.
Pulmonary vascular resistance | 15 weeks
  Change from baseline to 15 weeks, of pulmonary vascular resistance and total pulmonary resistance as measured during resting and exercise right heart catheterisation
Cardiac Output at rest and peak exercise | 15 weeks
  Change in cardiac output from baseline to 15 weeks as measured by right heart catheterisation at rest and on supine exercise
Change in resting and peak exercise mixed venous oxygen saturation | 15 weeks
  Change in mixed venous oxygen saturation from baseline to week 15, as measured from the central pulmonary artery during resting and exercise right heart catheterisation.
Left ventricular ejection fraction | 15 weeks
  Left ventricular ejection fraction as measured by cardiac MRI - change from baseline to 15 weeks following exercise therapy

OTHER OUTCOMES:
Profile of inflammatory cytokines | 15 weeks
  change in profile of pro-inflammatory serum cytokines as measured by multiplex ELISA from baseline to 15 weeks following exercise training.
Insulin resistance | 15 weeks
  Change in HOMA-IR score from baseline to 15 weeks following exercise therapy (scored from fasting serum c-peptide and glucose)

CONTACTS AND LOCATIONS:
Locations (1):
- Dr Martin Johnson, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: No